CLINICAL TRIAL: NCT06322407
Title: A Prospective, Randomized, Controlled, Blinded-endpoint Study to Evaluate the Efficacy and Safety of Stellate Ganglion Block for CM Treatment
Brief Title: Ultrasound-guided Stellate Ganglion Block for Treatment of Chronic Migraine in Adult
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Day surgery and Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2023-263-03-02
Record Dates: First submitted 2024-03-11; First posted 2024-03-21 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Chronic Migraine
Keywords: Chronic Migraine; Stellate Ganglion Block
MeSH Terms: interventions — Topiramate; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion Block plus standardized drug treatment group (Experimental): Besides orally topiramate plus ibuprofen as standardized drug treatment, patients will also receive SGBs plus standardized drug therapy; SGB will be performed once a week for 4 consecutive times in an individual series. The interval of each separate SGB procedure is 1 week. Every time patients with bilateral headache will be administered SGB alternately on each side at an interval of 40 min, and patients with unilateral headache will be administered SGB on the ipsilateral side;
  Interventions: Procedure: Stellate Ganglion Block (SGB); Drug: standardized drug treatment
- standardized drug treatment group (Active Comparator): The patients will only receive Topiramate plus ibuprofen as standardized drug treatment according to the guidelines for the treatment of CM.
  Interventions: Drug: standardized drug treatment

INTERVENTIONS:
Procedure: Stellate Ganglion Block (SGB) — All SGB procedures will be performed by the same experienced physicians. Patients will be positioned in a supine position with the neck slightly hyperextended and receive a SGB procedure using the B-ultrasound visualization technique (Aurora A5 Ultrasound, Risco Tech Co., Ltd.). 1% lidocaine 5mL (Shanxi Jinxin Shuanghe Pharm Co., Ltd.) will be injected below the prevertebral fascia on the surface of longus colli muscle
  Other Names: Ultrasound-guided Stellate Ganglion Block (SGB)
  Arms: Stellate Ganglion Block plus standardized drug treatment group
Drug: standardized drug treatment — Topiramate(Topiramate, Xi'an Yangsen Pharmaceutical Co., Ltd) will be started at a low dose and then increased gradually until optimally effective, side effects become intolerable, or the maximum recommended dose is reached. During the 4-week up-titration phase, the intention will increase dose weekly in 25 mg increments with the aim of reaching 50-100 mg/day. Ibuprofen((Fenbid, Tianjin Shike Pharmaceutical Co., Ltd)will be chosen as acute treatment, but no more than 10 times per month to avoid medication overuse headache.
  Other Names: topiramate plus ibuprofen

SUMMARY:
To assess the 6-months effects and safety of stellate ganglion block(SGB) for Chronic Migraine (CM) patients who failure to undergo preventive therapy and are seeking a more suitable non-pharmacological therapy.

DETAILED DESCRIPTION:
The investigators aim to investigate whether the stellate ganglion block(SGB) is better than traditional medication treatment and provides medical evidence for the clinical application and promotion of SGB to provide a minimally invasive, safe, and effective treatment for patients with chronic migraine(CM) who failed to receive standardized drug treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65 years;
2. Diagnosed with CM according to the International Classification of Headache Disorders, 3rd (ICHD-3) criteria [Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018;38:1-211].
3. not received prior prophylactic migraine treatment or, due to lack of efficacy or tolerability, had failed or had not been suitable for up to three previous prophylactic treatments from the following: Metoprolol/propranolol, amitriptyline, and flunarizine.

Exclusion Criteria:

1. BMI <15 kg/m2 or >35 kg/m2；
2. Previous SGB treatment；
3. History of other neurological disorders；
4. History of severe cardiopulmonary, hepatic or renal dysfunction；
5. History of allergies to any of the study drugs；
6. Patients with chronic use of opioids；
7. Preoperative coagulation abnormalities (activated partial thromboplastin time greater than 1.5 time normal value)；
8. Infection or mass near the puncture site；
9. Neck anatomic structural changes (caused by radiotherapy or surgery);
10. Pregnant or breast feeding;
11. Psychological disorders;
12. Refusal to sign informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
the change from baseline in mean monthly migraine days | 6-month period
  The primary outcome is the change from baseline in mean monthly (defined as 4 weeks) migraine days across 6-months follow-up period, which will be assessed by a blinded independent central review (BICR). Baseline is defined as the number of migraine days during the last 28 days prior to the randomization date. A migraine day is defined as a calendar day with symptoms of a migraine attack lasting at least 30 min.

SECONDARY OUTCOMES:
Proportion of patients achieved≥50% reduction in monthly migraine days | 1 month, 2 months, 3 months, 4 month，5 month and 6 month after surgery
  Proportion of patients achieved≥50% reduction
Total effective rate | 1 month, 2 months, 3 months, 4 month，5 month and 6 month after surgery
  Total effective rate = cure rate + markedly effective rate + effective rate
The mean Numeric Rating Scale(NRS) score during headache attack | at baseline, 1 month, 2 months, 3 months, 4 month，5 month and 6 month after surgery
  The Numeric Rating Scale(NRS) scoring method typically uses a score range of 0-10, with 0 indicating no pain or symptoms and 10 indicating the most severe pain or symptoms.
Patients satisfaction (PS) | 1 month, 2 months, 3 months, 4 month，5 month and 6 month after surgery
  Patients satisfaction (PS) evaluated by PS scores, which typically uses a score range of 0-10, with 0 indicating no patient satisfaction and 10 indicating the most patient satisfaction.
The six item headache impact test (HIT-6) | at baseline, 1 month, 2 months, 3 months, 4 month，5 month and 6 month after surgery
  The six item headache impact test (HIT-6) is a self-reported questionnaire measuring the "impact that headaches have on the ability to function on the job, at school, at home, and in social situations.
the Migraine Disability Assessment score(MIDAS) | at baseline, 1 month, 2 months, 3 months, 4 month，5 month and 6 month after surgery
  MIDAS is a reliable and validated scale measuring migraine-related disability regarding the need for medical care.. Higher MIDAS scores indicate more days with disability
The Pittsburgh Sleep Quality Index (PSQI) | at baseline, 1 month, 2 months, 3 months, 4 month，5 month and 6 month after surgery
  PSQI is a self-administered assessment of sleep disturbances that may affect sleep quality, including sleep apnoea, with a higher score indicating more severe sleep disturbances.
adverse events | at 0 day , 1 week, 2 week, 3 week, 1 month, 2 months, 3 months, 4 month，5 month and 6 month after surgery
  Proportion of participants with adverse events (AEs) and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
not yet decided